CLINICAL TRIAL: NCT01314183
Title: Enhancing the Effectiveness of Physical Therapy for People With Knee
Brief Title: Enhancing the Effectiveness of Physical Therapy for People With Knee Osteoarthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, g. kelly fitzgerald, Professor, Department of Physical Therapy, University of Pittsburgh, Agency for Healthcare Research and Quality (AHRQ)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01HS019624-01 (AHRQ)
Record Dates: First submitted 2011-02-23; First posted 2011-03-14 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis
Keywords: Knee; Physical Therapy; Exercise
MeSH Terms: conditions — Osteoarthritis; Motor Activity | interventions — Exercise; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- exercise (Active Comparator): Subjects in this arm receive 12 exercise sessions in 9 weeks.
  Interventions: Other: Exercise
- exercise + manual therapy (Active Comparator): Subjects in this group receive exercise combined with manual therapy techniques for 12 sessions in 9 weeks.
  Interventions: Other: Exercise; Other: manual therapy
- exercise + booster (Experimental): subjects in this arm will receive exercise sessions delivered with booster sessions (8 sessions in the first 9 weeks, 2 sessions at 5 months, 1 session at 8 months, and 1 session at 11 months).
  Interventions: Other: Exercise
- exercise + manual therapy + booster (Experimental): Subjects in this arm will receive exercise combined with manual therapy techniques and booster sessions.
  Interventions: Other: Exercise; Other: manual therapy

INTERVENTIONS:
Other: Exercise — The program starts with a 10 minute aerobic exercise warm-up (treadmill walking or stationary cycling). Subjects then perform a series of strengthening, stretching, and neuromuscular control activities which are core exercises for the program and mandatory. In addition to the above core exercises, therapists have the option to select additional optional exercise activities, based on the initial examination findings. These exercises will address strength or flexibility in the hip, and ankle if impairments are identified in the initial examination.
Other: manual therapy — The manual therapy (MT)techniques are maneuvers that are applied with manual force from the treating therapist. The MT techniques will include a series of accessory motion techniques, manual stretching , and soft tissue manipulation (deep massage to muscles and connective tissues associated with knee function). Core techniques include anterior-posterior and posterior-anterior tibiofemoral translations, superior-inferior and medial-lateral patellofemoral mobilizations, knee flexion and extension mobilizations that may be combined with varus-valgus stresses,medial-lateral tibial rotations, manual stretching of the quadriceps, rectus femoris, hamstring, and gastrocnemius muscles, and soft tissue manipulations of the quadriceps, peri-patellar tissues, hamstring, hip adductors, and gastroc-soleus muscle groups. There are optional MT techniques for the hip, and foot and ankle joints that can be selected by the therapist based on initial examination findings.
  Arms: exercise + manual therapy; exercise + manual therapy + booster

SUMMARY:
The overall aim of the project is to examine the clinical and cost-effectiveness of utilizing booster sessions(periodic face-to-face follow-up appointments that take place several weeks or months following discharge from the supervised therapy program designed to review the patient's current rehabilitation program, troubleshoot any problems with the program, and make recommendations for program progression or modification) in the delivery of exercise therapy, and supplementing exercise therapy with manual therapy techniques(manually applied treatment techniques such as joint mobilization/manipulation, manual traction, soft tissue manipulations, passive stretching and range of motion). The investigators will do this in a randomized, multi-center, clinical trial. The investigators hypothesize that adding manual therapy techniques will be more clinically effective than exercise alone and that using booster sessions will maintain longer term clinical effects and be more cost-effective than not using booster sessions.

DETAILED DESCRIPTION:
Exercise therapy (ET) is effective as the first line of treatment for reducing pain and disability in patients with knee osteoarthritis (OA), but studies show its effects diminish considerably over time. 'Booster' intervention sessions (periodic face-to-face follow-up appointments following discharge from supervised therapy designed to review and progress the patient's home program, troubleshoot problems with the program, etc.) have been recommended to make beneficial effects endure however this recommendation has not been adequately tested. There are also indications that manual therapy (MT), manually applied treatment techniques such as joint mobilization/manipulation, manual traction, soft tissue manipulations, and passive stretching, when combined with ET, may improve the overall effectiveness of rehabilitation for reducing pain and disability, and, may significantly delay or reduce the need for total knee arthroplastic surgery and reduce medication intake in people with knee OA. However, current published evidence-based treatment guidelines indicate there is not enough data to make a definitive recommendation regarding the use of MT with ET in rehabilitation programs. Therefore, the overall aim of the project is to examine the clinical and cost-effectiveness of utilizing booster sessions in the delivery of ET, and supplementing ET with MT techniques.The study will be a multi-center,randomized clinical trial, using a 2 x 2 factorial design (factor 1 = booster vs no booster, factor 2 = ET alone vs ET + MT). Three hundred subjects (100 per study site) with knee OA will be randomized to one of the following groups: 1) ET - no booster, 2) ET - with booster, 3) MT + ET - no booster sessions, 4) MT + ET - with booster sessions. Clinical outcome measures (WOMAC, knee pain, global rating of change and performance-based measures of function) will be taken at baseline (prior to randomization), at the completion of the initial therapy sessions (9 weeks) and at 1 year follow-up. The primary endpoint for clinical outcome will be the WOMAC at 1 year.For the cost effectiveness analysis, the primary cost outcome will be osteoarthritis treatment costs from the societal perspective, which will include health system costs for implementing each intervention, medical/surgical costs (primary, secondary, and tertiary care costs), and personal costs to participants (travel, non-funded medications, time off work, and quality-of-life burdens). The primary effectiveness outcome measure will be quality-adjusted life-years (QALYs), derived using quality of life utilities from EQ-5D scores. Cost and effectiveness values between interventions will be compared via incremental cost-effectiveness ratios, yielding incremental costs per QALY gained when a given intervention is chosen. Secondary analyses will examine cost-effectiveness from health system and from patient perspectives. Cost and effectiveness data will be obtained at 1 year and 2 year follow-ups. The 2 year follow-up will be the primary endpoint for the cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older
* Meet the American College of Rheumatology (ACR) clinical criteria for a diagnosis of knee OA. The ACR clinical criteria for knee OA includes knee pain plus 3 of the following 6 criteria:
* age > 50 years,
* morning stiffness of < 30 minutes,
* crepitus on active movement,
* tenderness of the bony margins of the joint,
* bony enlargement of the joint noted on exam,
* lack of palpable warmth of the synovium. Based on this criteria, a subject who is less than 50 years but has knee pain and 3 of the other 5 criteria would also be classified as having knee OA.

Exclusion Criteria:

* do not meet the ACR clinical criteria for knee OA,
* are scheduled for total knee arthroplasty (TKA) surgery,
* have undergone TJA surgery on any lower extremity joint,
* exhibit uncontrolled hypertension (i.e. individuals not currently taking medication for hypertension whose systolic blood pressure is greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg at rest),
* have complaints of low back pain or other lower extremity joint pain that affects function at the time of recruitment,
* have a history of neurological disorders that would affect lower extremity function (stroke, peripheral neuropathy, parkinson's disease, multiple sclerosis, etc.),
* are women who are pregnant.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Change from baseline at 9 weeks, 1 year and 2 years
  Self report measure of pain, stiffness, and physical function for people with knee osteoarthritis.

SECONDARY OUTCOMES:
Cost/Utility Ratio | 2 years
  In the analysis, the effectiveness term will be quality adjusted life years, which is the product of the quality of life utility associated with a health state and the length of time lived in that state, summed over time. Utilities are a measure of preference for a health state and range from 0 (death) to 1 (perfect health). In this analysis, utilities will be derived from EQ-5D scores. The cost-effectiveness ratio (or, in this analysis, the cost-utility ratio) is the difference in cost divided by the difference in quality-adjusted life-years between intervention groups.
Change in Numeric Knee Pain Rating Scale | Change from Baseline to 9 weeks, 1 and 2 years
  Subjects will rate their worst knee pain in the last 24 hours using an 11 point numeric pain rating scale with 0 representing "no pain" and 10 representing " the worst pain imaginable."
Global Rating of Change | Change from baseline to 9 weeks, 1 and 2 years
  The global rating of change is a 15 item scale in which subjects will rate the degree to which their knee condition has changed from the time treatment was initiated to the present.24 The subject responds to the following query: "Please rate your overall knee's condition from the time you began treatment until now (check only one)." The items range from "A very great deal better" to "A very great deal worse."
Change in Timed Up and Go Test Time | Change from Baseline to 9 weeks and 1 year
  On the command "go" subjects will stand up from a chair, walk 3 meters, turn around, return to the chair and sit down. The time it takes to complete this task will be recorded.
Change in 30 second time chair rise test. | Change from Baseline to , 9 weeks, 1 year
  Subjects will be seated with their arms crossed in front of their chest. On the command "go" subjects will stand up and sit down for as many trials as they can in a 30 second period.
Change in Self-paced Walk Test Time | Change from Baseline to 9 weeks, 1 year
  Subjects will walk 4 lengths of a 10 meter indoor course in response to the instructions, "Walk as quickly as you can without overexerting yourself."
Change in Pain belief screening instrument | Change in Baseline to 1 year
  7 item instrument that queries the subject about their pain and how they believe pain limits or does not limit their ability to perform daily activities, social and liesure interactions, mood, etc.
Change in Beck Anxiety Index (BAI) | Change from Baseline to 1 year
  The BAI consists of 21 items, each item scored 0-3, with higher scores representing higher levels of anxiety.
Change in Center for Epidemiological Studies Depression Scale (CES-D) | Change from Baseline to 1year
  The CES-D is a 20-item self-report depression scale, each item scored 0-3, with higher scores representing greater symptoms of depression.
Change in EQ-5D | Change from Baseline to 1 and 2 years
  The EQ-5D is a generic health-related quality of life measure. The EQ-5D consists of the following five dimensions: 1) Mobility, 2) Self-care, 3) Usual activities, 4) Pain/discomfort, and 5) Anxiety/depression (AD).Each dimension has three possible levels (i.e., 1, 2, or 3), representing "no problems," "some problems," and "extreme problems," respectively. Respondents are asked to choose one level that reflects their "own health state today" for each of the five dimensions.
OARSI Responder Criteria | 9 weeks and 1 year
  Responder criteria included 1) greater than or equal to 50% improvement in WOMAC pain or WOMAC function and an absolute improvement of greater than or equal to 20, or 2) improvement in at least 2 of the following 3 scores: 20% improvement in pain and absolute change ≥ 10 on WOMAC pain score, 20% improvement in pain and absolute change ≥ 10 on WOMAC function score, or moderate or greater improvement (≤ 4) on a 15 point global rating of change scale.

CONTACTS AND LOCATIONS:
Overall Officials: G. Kelley Fitzgerald, PT, PhD, Principal Investigator — University of Pittsburgh; Julie M Fritz, PT, PhD, Principal Investigator — Intermountain Healthcare, Salt Lake City, UT; John D Childs, PT, PhD, Principal Investigator — Army-Baylor University, San Antonio, TX; J. Haxby Abbott, PT, PhD, Principal Investigator — University of Otago, Dunedin, New Zealand
Locations (3):
- United States (3):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Army-Baylor University, San Antonio, Texas
  - Intermountain Healthcare, Salt Lake City, Utah

REFERENCES:
- [Derived] Bove AM, Smith KJ, Bise CG, Fritz JM, Childs JD, Brennan GP, Abbott JH, Fitzgerald GK. Exercise, Manual Therapy, and Booster Sessions in Knee Osteoarthritis: Cost-Effectiveness Analysis From a Multicenter Randomized Controlled Trial. Phys Ther. 2018 Jan 1;98(1):16-27. doi: 10.1093/ptj/pzx104. PMID 29088393
- [Derived] Fitzgerald GK, Fritz JM, Childs JD, Brennan GP, Talisa V, Gil AB, Neilson BD, Abbott JH. Exercise, manual therapy, and use of booster sessions in physical therapy for knee osteoarthritis: a multi-center, factorial randomized clinical trial. Osteoarthritis Cartilage. 2016 Aug;24(8):1340-9. doi: 10.1016/j.joca.2016.03.001. Epub 2016 Mar 10. PMID 26973326